CLINICAL TRIAL: NCT05978947
Title: Effect of Sperm Preparation by a Microfluidic Chip Method Versus a Density Gradient Centrifugation Method on Semen Parameters
Brief Title: Microfluidic Chip Method Versus Density Gradient Centrifugation Method on Semen Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Ernest Hung-Yu Ng (Other)
Responsible Party: Sponsor-Investigator, Professor Ernest Hung-Yu Ng, Clinical Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 23-233
Record Dates: First submitted 2023-06-29; First posted 2023-08-07 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Infertility
Keywords: Semen parameters; Microfluidic chip; Density Gradient Centrifugation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial aims compare the effect of sperm preparation by a microfluidic chip method versus a density gradient centrifugation method on semen parameters prior to the start of a randomized trial comparing the effects of the two sperm preparation methods on the cumulative live birth rates of in vitro fertilization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the laboratory staff in the IVF laboratory performing sperm preparation will be aware of the group assignment. Another laboratory staff who is not involved in performing sperm preparation and is not aware of the group assignment will perform the semen analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Microfluidic Chip Method (Experimental): The Sperm Separation Device - ZyMōt Multi 850µL device (ZyMōt Fertility, Inc) will be used. The microfluidic chamber will be used based on the manufacturer's instructions. 850 μL of the semen sample will be added to the inlet port of the device and 750 μL of fertilization media will be added to the outlet port. The device will then be incubated in 6% CO2 at 37°C. After 30 minutes, 500 μL of the prepared sample at the outlet port will be removed and pipetted into a labelled test tube. The final volume will be adjusted to 1mL for sperm counting.
  Interventions: Device: ZyMōt Multi 850µL device
- Density Gradient Centrifugation Method (Active Comparator): After liquefaction, sperm preparation will be completed by a discontinuous density gradient centrifugation method, using Pureception (CooperSurgical, Denmark) sperm density gradient media. The resulting sperm pellet after centrifugation will be washed once with the sperm washing medium (G-IVF Plus, Vitrolife, Sweden) The washed spermatozoa will be resuspended with the same medium, adjusting the final volume to 500 μL. The final volume will be adjusted to 1mL for sperm counting.
  Interventions: Device: Density Gradient Centrifugation Method

INTERVENTIONS:
Device: ZyMōt Multi 850µL device — The ZyMōt Multi 850µL device is a laboratory tool designed for use in assisted reproductive technology (ART) procedures such as intrauterine insemination (IUI) and in vitro fertilization (IVF). It is a sperm preparation device that uses a proprietary patented technology to isolate and select motile sperm from semen samples for use in ART procedures.
  Arms: Microfluidic Chip Method
Device: Density Gradient Centrifugation Method — Density gradient centrifugation is a laboratory technique used to separate and isolate different types of cells or particles based on their density. It is commonly used in various applications, including cell biology, immunology, and assisted reproductive technology (ART).
  Arms: Density Gradient Centrifugation Method

SUMMARY:
Infertility affects many couples, with male infertility being a common cause. In vitro fertilization (IVF) is an effective treatment, but its success rates are not high. Semen quality can affect IVF outcomes, and the current method used to process semen can damage the sperm and DNA. Scientists are now testing a new method called microfluidic chip technology, which reduces DNA damage and increases sperm movement. This study will compare the effectiveness of the chip method and the current method on semen quality in men attending a fertility clinic. The study will randomly assign semen collected to one of the two methods and assess the semen quality using different tests, as well as the difference in using two different microfluidic chip platform . The primary outcome will be DNA fragmentation, and other outcomes include sperm count and motility. Semen samples would be collected from study subjects for analysis and that both the samples and results would not be used in patients' treatment.

DETAILED DESCRIPTION:
Infertility affects one in six couples and is getting more common as many women delay marriage and childbirth for various reasons. In vitro fertilization (IVF) is the most effective treatment for couples with long standing infertility and has treated millions of infertile couples over the world since the first birth of IVF was reported more than 40 years ago. However, despite advances in technology, the pregnancy and birth rates remain around 35% and 25% per transfer in Europe in 2018. Among all infertile couples, 20-30% are due to male infertility. Semen parameters may affect the IVF outcomes and it was hypothesized that the relative contribution of sperm to a live birth is around 10-15%.

IVF involves hormone injections to stimulate a woman's ovaries to produce a number of oocytes which are collected by a minor operation and then mixed with sperm to form embryos in the laboratory. Usually, one or two embryos are transferred to the uterus 2-5 days after oocyte retrieval. In IVF, semen samples produced by husbands are commonly processed by a density gradient centrifugation method to isolate the better spermatozoa for fertilization. The density gradient centrifugation can enrich spermatozoa with relatively good motility and normal morphology. It is possible to recover spermatozoa from semen specimens with a very low sperm density. It can provide a relatively good yield. However, it requires technical training to set up the density gradient consisting of two media with different densities. During semen processing, spermatozoa are centrifuged through the gradient. It is known that centrifugation causes considerable damage to spermatozoa by the reactive oxygen species produced during the process. Reactive oxygen species are known to be one of the major causes leading to sperm DNA fragmentation and subsequent adverse outcomes including implantation failure and miscarriage. A meta-analysis showed sperm DNA damage has a negative effect on clinical pregnancy following IVF.

A microfluidic chip, which is a miniaturized device containing channels and chambers in the microscale range for nanoparticle preparation, is being used as an alternative sperm preparation technique recently. By employing microfluidic technology, spermatozoa can go through the chip that closely simulates the natural selection in the female genital tract microenvironment. The technology enables the selection of high-quality motile spermatozoa from semen samples without the need for centrifugation, leading to reduced reactive oxygen species formation.

Studies have consistently demonstrated that the use of a microfluidic chip method greatly reduces DNA fragmentation and increases motility when compared with the density gradient centrifugation method.

This randomized controlled trial aims compare the effect of sperm preparation by a microfluidic chip method versus a density gradient centrifugation method on semen parameters prior to the start of a randomized trial comparing the effects of the two sperm preparation methods on the cumulative live birth rates of in vitro fertilization.

Objectives:

The first objective of this randomized controlled trial is to compare the effect of sperm preparation by a microfluidic chip method versus a density gradient centrifugation on semen parameters. The hypothesis is that the use of sperm preparation by a microfluidic chip method improves semen parameters.

The second objective is to compare the effect of two different microfluidic chip platforms on semen parameters.

Trial design:

Men attending at the Centre of Assisted Reproduction and Embryology, Queen Mary Hospital for fertility treatment will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Sperm concentration of the raw semen with at least 5 million motile sperm per ml with a total volume of not less than 1.5ml.

Exclusion Criteria:

* Sperm concentration of the raw semen of less than 5 million motile sperm per ml
* Men unable to provide an ejaculated semen sample

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
DNA fragmentation by Comet assay | 1 months
  Measurement of DNA fragmentation by Comet assay using the Olive tail moment as the quantitative metric.

SECONDARY OUTCOMES:
Sperm count | 1 months
  Sperm count
Forward motility | 1 months
  Assessment of forward motility of sperm by manual observation using the World Health Organization (WHO) criteria.
Sperm velocities measured by CASA | 1 months
  Quantitative analysis of sperm velocities using computer-assisted sperm analysis (CASA) system, including assessment of forward motility, curvilinear velocity, and linearity.
Morphology | 1 months
  Quantitative assessment of sperm morphology by manual observation using the Tygerberg strict criteria.
Sperm aneuploidy | 1 months
  Quantitative measurement of sperm aneuploidy by fluorescence in situ hybridization (FISH) using probes for chromosomes X, Y, 13, 18, and 21.
Calcium ionophore A23187 -induced acrosome reaction assay | 1 months
  Quantitative measurement of acrosome reaction in sperm induced by calcium ionophore A23187 using flow cytometry.
Artificial intelligence analysis | 1 months
  Quantitative analysis of sperm morphology using artificial intelligence algorithms.
Intact oocyte/hemizona binding assay | 1 months
  Quantitative measurement of sperm binding to intact oocytes or hemizona using the intact oocyte/hemizona binding assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No